CLINICAL TRIAL: NCT04710381
Title: Pilot, Monocentric, Phase-IV Clinical Trial Assessing the Clinical Effect of Peroral Immunomodulation Treatment Using the IMUNOR® Preparation in the Prevention of COVID-19 Disease
Brief Title: IMUNOR® Preparation in the Prevention of COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FNO-IMUNOR-2020
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: Covid19; prevention; pork dialyzed leukocyte extract; immunomodulation
MeSH Terms: conditions — COVID-19 | interventions — IMUNOR

STUDY DESIGN:
Intervention Model Description: The study treatment (IMUNOR) will be administered to one group of study subjects only.
Masking Description: No masking will be used in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMUNOR (Experimental): Study subjects in this arm will receive IMUNOR preparation as prevention against COVID-19 disease.
  Interventions: Drug: IMUNOR

INTERVENTIONS:
Drug: IMUNOR — The intervention consists of the administration of IMUNOR as prevention against COVID-19 disease

SUMMARY:
The aim of the study is to achieve prevention of COVID-19 disease in healthcare professionals with the administration of the IMUNOR® preparation, and decreasing the symptoms should the disease appear.

DETAILED DESCRIPTION:
This prospective study is designed to collect data for evaluation of the preventive and therapeutic effect of the IMUNOR® preparation, which is commonly used to treat patients with laboratory or clinical manifestations of immunity disorders. Administration of immunomodulation treatment will be based upon a willing informed consent with the administration of the drug and based upon random selection. The study subjects will receive IMUNOR® preventively; the anticipated preventive effect when using one packing (4 vials) is 6 weeks, and 12 weeks when using two packings. Should any signs of acute illness appear (increased body temperature, cough, loss of smell and taste, etc.), a treatment dose of IMUNOR®, i.e. 1 vial/day (total of 4 vials) will be administered immediately. Monitoring of individual patients will take 6 weeks (1 packing) or 12 weeks (2 packings) from the beginning of IMUNOR® administration. The clinical condition of study subjects will be monitored on a daily basis. At the same time, the possible onset of symptoms will be recorded.

The obtained data will be compared with a control group consisting of patients followed by the Department of Preventive Medicine, University Hospital Ostrava.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects 18-60 years old
* Ability to cooperate upon the study and to give informed consent

Exclusion Criteria:

* Use of any other immunomodulation treatment one month prior to enrolment and in the course of the study
* Acute disease of the cardiovascular, urogenital, respiratory or nervous system

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Prevention of COVID-19 disease | 6 or 12 weeks
  The incidence of COVID-19 disease among the studied population will be assessed.
Prevention of hospitalisations due to COVID-19 | 6 or 12 weeks
  The number of study subjects requiring hospitalisation due to COVID-19 will be observed

SECONDARY OUTCOMES:
Incidence of sick-leave episodes | 6 or 12 weeks
  The number of study subjects requiring a sick-leave due to COVID-19 will be observed

CONTACTS AND LOCATIONS:
Overall Officials: Jaromír Bystroň, Ass.Prof.,MD,CSc., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.